CLINICAL TRIAL: NCT03010124
Title: Prognostic and Predictive Biomarkers in Ovarian Cancers
Acronym: OvBIOMark
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A01183-46; 2015/2290 (Other: CSET number)
Record Dates: First submitted 2016-12-13; First posted 2017-01-04 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with ovarian cancer (Other)
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample

SUMMARY:
The investigators therefore propose to conduct a biological study of prospectively collected patient tumour samples, ascites, blood and other residual samples (feces, urine, vaginal smear) throughout the disease course where markers (at diagnosis and their change with treatment) will be correlated to outcome in order to investigate how genetic diversity in OC prior to treatment and adaptation following treatment contribute to chemotherapy resistance. In addition freshly collected ascitic samples (and tumour samples) will be subjected to ex vivo DNA repair functional assays and isolated in primary culture (and established as xenografts) for target validation experiments.

ELIGIBILITY:
Inclusion Criteria:

1. New patient with a diagnosis of OC, or
2. Previously treated patient with frozen or formalin fixed paraffin embedded primary tumour sample available that can be retrieved by the center presenting with progressive disease, and consenting to CT guided biopsy of relapsed disease, or
3. Previously treated patient with frozen or formalin fixed paraffin embedded primary tumour sample available that can be retrieved by the center scheduled for surgery for relapsed disease.
4. Signed informed consent
5. Age ≥ 18
6. Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

1. Patients who do not fit the inclusion criteria and those who refuse an antitumoral treatment;
2. Coagulation abnormalities that contra-indicates the biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-09-26 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Correlation of baseline biomarkers with PFS will occur at 12 months following last patient inclusion
  up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No